# Annexure 1

# Data Analysis Plan (Samvedana Plus)

The group should prepare the data analysis plan and share

| Proposed title | The effectiveness of a multi-level intervention to reduce violence and increase condom use in intimate partnerships of sex workers in Karnataka: findings from a clustered randomised controlled trial |
|---|---|
| Journal options | 1. Lancet Global Health (17.7) |
| Note journal, impact factor and word limit | 2. American Journal of Public Health |
| , , , | (3.86) |
| | 3. Social Science Medicine (2.8) |
| Proposed lead authorship | First joint author: |
| Define lead authors names, organisations and role in | Shajy Isac and Lucy Platt will conduct the |
| authorship | analysis and prepare the draft together |
| (i.e. who will conduct analyses, who will write first | Second: Prakash Javalkar will support the |
| draft) | analysis and partial draft write-up |
| , | Last: |
| | Lori will review the analysis and the first draft |
| | of manuscript |
| Potential additional authors (who may be invited to | Co-authors from KHPT, LSHTM, and UoM to be |
| join) | decided. Sequencing will be decided based on |
| Name/Organisation | the contribution of the co-authors. Rachel |
| | Jewkes to be invited as co-author |
| Proposed Research Question | What is the effect of the Samvedena Plus |
| Note if this is a primary or secondary study question | intervention on reducing violence and |
| | increasing condom use within intimate partner |
| | relationships among female sex workers in |
| | Karnataka? |
| Define data to be used in the analysis | Quantitative data collected through face-to- |
| <ul> <li>Quantitative data plans should detail all</li> </ul> | face interview with female sex workers would |
| dependent and independent variables (including | be used to analyze the above-stated research |
| categorisation of variables) | questions. |
| <ul> <li>Qualitative data plans should detail data themes</li> </ul> | 4.55.5.5. |
| - Quantative data plans should detail data themes | The table below summarises the definitions of |
| | indicators, the questions to be used for |
| | analysis and the source of information. |
| <b>Table.</b> Indicators, analytical variables and data source f | |

**Table.** Indicators, analytical variables and data source for primary and secondary outcomes

| Research question # | Indicator(s) | Variable | Source of information | Survey data round | Analysis |
|---|---|---|---|---|---|
| 1. Primary ou | tcome | | | | |
| What is the | 1. Proportion of | <b>Q901(e to m):</b> How | Individual | End-line data | Comparison |
| effect of the | FSWs who | often experienced | FTFI | | of responses |







| Samvedena<br>Plus<br>intervention<br>on reducing<br>violence and<br>increasing<br>condom use<br>within<br>intimate | report physical o sexual violence from intimate partners in the past 6 months. | from intimate partner-1 (coded >0 in any of violence act from e to m) | (Responses<br>for IP1 that<br>is most<br>significant<br>partner) | | between<br>intervention<br>and control<br>arms |
|---|---|---|---|---|---|
| partner<br>relationships<br>among<br>female sex<br>workers in<br>Karnataka? | 2. Proportion of FSWs experience severe physical and/or sexual violence from intimate partners in the past 6 months | often experienced each act of violence in last 6 months from intimate partner-1 (Coded as 3 in any of e to f and/or coded>0 in any of g to m) | Individual<br>FTFI<br>(Responses<br>for IP1 that<br>is most<br>significant<br>partner) | End-line data | Same as above |
| | 3. Proportion of FSWs we report consisten condom use in their intimate relationsh within the past 30 days. | who how often are condoms (either male or female) used while having sexual intercourse with this partner? Would you say every time, most of the | Individual<br>FTFI<br>(Responses<br>for IP1 that<br>is most<br>significant<br>partner) | End-line data | Same as above |







| T | | | Ι | | 1 | <del> </del> |
|---|---|---|---|---|---|---|
| | | | sensitivity analysis | | | |
| | | | removing any | | | |
| | | | individuals not | | | |
| | | | reporting sex in the | | | |
| | | | last 30 days from the | | | |
| | | | analysis. | | | |
| 2. Secondary of | out | comes | | | | |
| | 4. | Reduced | Increase in % of | Individual | Endline | Comparison |
| | | acceptance | FSWs who said all of | FTFI | | of responses |
| | | of violence | the following | | | between |
| | | by their IPs | actions were not | | | intervention |
| | | | acceptable or | | | and control |
| | | | justified (composite | | | arms |
| | | | variable) : | | | |
| | | | <b>Q801:</b> Do you think | | | |
| | | | it is acceptable if a | | | |
| | | | man beats his lover | | | |
| | | | if she has done | | | |
| | | | nothing wrong? | | | |
| | | | <b>Q802:</b> Is a man | | | |
| | | | justified if he beats | | | |
| | | | her if she does not | | | |
| | | | prepare his food | | | |
| | | | well or on time? | | | |
| | | | Q803: Is a man | | | |
| | | | justified to beat her | | | |
| | | | if she continues to | | | |
| | | | see clients when he | | | |
| | | | has asked her not | | | |
| | | | to? | | | |
| | | | <b>Q804:</b> Is a man | | | |
| | | | justified to beat her | | | |
| | | | if she refuses to | | | |
| | | | have sex with him | | | |
| | | | on a particular | | | |
| | | | night? | | | |
| | | | <b>Q805:</b> Is a man | | | |
| | | | justified to beat her | | | |
| | | | if she goes out | | | |
| | | | without his | | | |
| | | | permission? | | | |
| | | | <b>Q807:</b> Is a man | | | |
| | | | justified in beating | | | |
| | | | his lover if he fails to | | | |
| | | | provide for her | | | |
| | | | financially? | | | |
| 1 | | | · · · | L | 1 | 1 — |







| | | Q808: Is a man justified in beating his lover if he has multiple lovers? | | | |
|---|---|---|---|---|---|
| 5 | disclosure of<br>IPV | Increase in % of FSWS reporting incidence of violence to the following individuals: Q903 (a to x): Who, if anyone, have you told about the violence you experienced from you IP? (Denominator = those who've experienced any sexual/physical violence in last 6 months (response y); Numerator = responses a to x) | Individual<br>FTFI | Endline | Comparison of responses between intervention and control arms |
| 6 | 6. Increased knowledge of self-protection strategies | Increase in % FSWs who have reported protection strategies: a) identifying allies; or b) identifying individual counter measures. Q1223: Have you ever developed a safety plan to prevent violence from your intimate partner? | Individual<br>FTFI | Endline | Same as above |
| 7 | 7. Increased self-efficacy to negotiate condom use with IP | Increase in % FSWs reporting fully confident (response 3) to Q712: How confident are you that you can persuade your intimate partner(s) | Individual<br>FTFI | Endline | Same as above |







| | | to use condom in future? | | | |
|---|---|---|---|---|---|
| 8 | 8. Increased solidarity among FSWs around issues of IPV | Increase in % FSWs reporting always/most of times to either: Q1001: Can you confide in other sex workers if you need to talk about your problems with intimate partners? OR Q1002: Can you go to your fellow sex workers for help at times of intimate partner? | Individual<br>FTFI | Endline | Same as above |

Data collection: BL [Jul-Aug'14]; ML [Aug, Oct-Dec'16]; EL [Jul-Sep'17]

**Intervention:** April 2015 to Jun-2017

# A priori confounders for primary outcomes

#### Individual- level

- Age (Q301: how old are you?)
- Literacy (Q302: can you read and write)
- Duration of sex work (Q402: how old were you when you started sex work MINUS Q301: how old are you?)
- Income other than sex work/Total income (Q310: what is your average monthly income from any activities other than sex work? /Q310 PLUS Q311: what is your average monthly income from sex work)
- Place of solicitation (Q403: Where do you generally solicit/pickup most of your clients?)
- Number of sex work clients (Q405: How many clients do you have sexual intercourse in a typical week?)
- Number of intimate partners -> (Q501: How many main/intimate (regular) partners do you currently have?)
- Intimate Partner caste -> caste difference (Q511: what is the caste or tribe of this partner? AND Q306: what is your caste or tribe?)
- Intimate Partner age difference? (Q506: what is the current age of this partner? AND Q301: how old are you?)
- Intimate Partner frequency of visit (Q514: how often does this partner visit you?)
- Number of children (Yes/No) Total (with intimate partner + others) (Q307: do you have children? If yes, how many?)







- Membership of Community Based Organisation (Q1204: are you member of any sex worker collective (CBO)?)
- Alcohol use (IP, FSW) (any + during sex) (Q533: how often does this IP come to you drunk or get drunk in your presence? OR Q534: during the past month, how often was this IP under the influence of alcohol when he had sex with you? AND Q535: during the past month, how often were you under the influence of alcohol when you had sex with this IP?

  AND Q414a: during the past month, have you consumed drinks containing alcohol? AND Q414b: during the past month how frequent did you get drunk?) For all these indicators we are referring to regular alcohol use (every time/often) as an indicator of heavy alcohol use for intimate partners (533, 534, 535). For FSW every day or at least once a week is heavy use. (414a and 414b)
- Intimate partner knowing sex work status (Q518: does this partner know about your sex work profession?)
- Practiced sex work outside the village (Q402c: In the last 12 months, have you ever practiced sex work anywhere other than the village where you live?)
- Moved away from the state/district (Q402d: Which were the different places where you had done sex work during the last 12 months?)
- Village and FSW population size strata

## Cluster-level confounders (taken from baseline dataset)

• Baseline levels of outcomes

### A priori confounders for secondary outcomes.

As above

## **Analysis methods**

- Quantitative data plans should detail statistical analysis methods
- Qualitative data plans should detail theoretical analysis methods

The primary outcome will be an adjusted, individual-level intention to treat analysis, comparing outcomes in interventions and control villages using end-line survey as the primary analysis for primary outcomes and secondary outcomes (see above). We will include all women surveyed at each time point (i.e. don't dismiss women who aren't captured at baseline)

The analysis will be conducted in two stages:

<u>Stage one: descriptive analysis (Figure 1 – Tables 1-2)</u>

We will check imbalance between confounders and socio-demographic indicators (see above) between arms within baseline data using blinded datasets and reporting proportions only to avoid deductive disclosure (since we have an imbalance in clusters between arms).







This comparison is just to observe differences. We will review the tables as a critical reader to assess imbalances making judgements on the importance of imbalances depending on their association with outcomes — i.e. bigger imbalances of something not strongly related to the outcome is less important than smaller imbalances of outcomes.

We will report cluster-level summaries (mean of the cluster-level means by Trial arm for each primary and secondary outcomes as a way of double checking our analyses and since risk differences are easier to interpret than odds ratios used in the individual level analysis. This is summarised in Table 2.

<u>Stage two: individual –level analysis with mixed</u> effects logistic model (Table 3)

As we have more than 20 clusters, we will conduct individual-level analysis with a mixed effects logistic model. We will fit dummy variables for strata (village population size-> 1-33 percentile; 34-67 percentile; 68-100 percentile; number of FSWs <=12 FSWs; > 12 FSWs). We will adjust for confounders in the following way:

- Outcome variables are adjusted for at a cluster level using mean <u>baseline summaries</u> (we need to check cluster sizes through – perhaps better to stratify if clusters are too small)
- Other variables will be adjusted for at individual level <u>using endline data</u>— only adjust for those variables that strongly predict outcome (a priori confounders but not on causal pathway) and where we think there is variability (drawing on descriptive analysis of baseline – stage 1).

For the covariates that were not measured at baseline (i.e. alcohol or mobility) we should check if they are on the causal pathway or if they were discussed in the intervention. We will not include them in the main analysis but conduct a sensitivity analysis.

Draft Data analysis plan: 23<sup>th</sup> October, 2017 Final Data analysis plan: 31<sup>st</sup> October, 2017

Timelines







| Note timelines for completion of each step in the writing process (add additional steps as appropriate) | Draft unblinding protocol: 23 <sup>rd</sup> October,2017 Data cleaning and basic coding: 10 <sup>th</sup> November, 2017 Draft analysis: By 2 <sup>nd</sup> December, 2017 Final analysis: 15 <sup>th</sup> January, 2018 First draft: End February'2018 Journal submission: End March'2018 |
|---|---|
| Review process If the authors request review of the data analysis plan by someone external to the writing team, note the name of the reviewer, timelines and document feedback. | Will this data analysis plan be reviewed? YES/NO Shajy, Mitzy, Lori, Parinita, Rachel, Tara |
| Changes If changes are subsequently suggested to the data analysis plan, detail the suggested changes and details of review and agreement by the authors and the reviewer (if relevant) | |
| Notes | |





